CLINICAL TRIAL: NCT03947346
Title: Biomarkers of Renal Dysfunction in Neuroblastoma Survivors
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 19-160
Record Dates: First submitted 2019-05-09; First posted 2019-05-13 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Neuroblastoma Survivors
Keywords: Kidney Function; Biomarkers; 19-160

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- survivors of neuroblastoma treated with nephrotoxic therapy: Upon enrollment, all subjects will receive a urine collection kit by mail. Participants will bring in a first-morning urine specimen on the day of their routinely scheduled long-term follow-up visit, and will then have an additional blood and urine sample drawn with their other clinical care labs upon arrival to MSK.
  Interventions: Other: Urine sample

INTERVENTIONS:
Other: Urine sample — The urine collected from the first morning void will be used to assess urine creatinine and microalbumin. The fresh urine specimen will be analyzed for novel urinary biomarkers of (urinary NGAL, TGF-β1, IL-18 and KIM-1). Serum BUN, creatinine, and cystatin-C will be assessed using serum samples drawn for routine clinical care.

SUMMARY:
The main purpose of this study is to learn more about biomarkers of kidney function in the blood and urine of neuroblastoma survivors. A biomarker is a biological molecule found in blood, urine, other body fluids, or tissues that is a sign of a normal or abnormal process, or of a condition or disease. A biomarker may be used to see how well the body responds to a treatment for a disease or condition.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of neuroblastoma between 0-18 years of age
* < 21 years of age at time of study enrollment
* Two or more years from completion of systemic chemotherapy and/or radiation therapy

Exclusion Criteria:

* Patients treated with observation only
* Patients with multiple primary cancers

Max Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Childhood cancer survivors followed by the Pediatric Long-Term Follow-Up (LTFU) Program will be recruited for the current study.
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2019-05-09 (Actual); Primary Completion 2025-07-15 (Actual); Study Completion 2025-07-15 (Actual)

PRIMARY OUTCOMES:
indicators of renal injury | 2 years
  urine collected from the first morning void will be used to assess urine creatinine

CONTACTS AND LOCATIONS:
Overall Officials: Danielle Friedman, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.
Supporting Information: SAP, ICF

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm